CLINICAL TRIAL: NCT01709474
Title: Vitamin D3 Effects on Immune Function in Pediatric Systemic Lupus Erythematosus (SLE)
Brief Title: Vitamin D3 Treatment in Pediatric Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow enrollment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ALE05
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Vitamin D3; Vitamin D deficiency; IFN alpha expression
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 6000 IU (Experimental): 6000 IU of vitamin D3 by mouth daily until the subject's serum 25(OH) level is ≥ 40ng/mL at which point the supplementation dose is reduced to 4,000 IU/day. Note: Subjects weighing <40 kilograms (kg) at study entry will receive their dose five days a week and all other subjects seven days a week.
  Interventions: Drug: Vitamin D3 6000 IU
- Vitamin D3 400 IU (Active Comparator): 400 IU/day of vitamin D3 by mouth daily.
  Interventions: Drug: Vitamin D3 400 IU

INTERVENTIONS:
Drug: Vitamin D3 6000 IU — Subjects will receive 6,000 IU of vitamin D3 by mouth daily until the subject's serum 25(OH) level is ≥ 40ng/mL at which point the supplementation dose will be reduced to 4,000 IU/day. Note: Subjects weighing <40 kilograms (kg) at study entry will receive their dose five days a week and all other subjects seven days a week.
  Other Names: high-dose vitamin D; high-dose cholecalciferol (D3); high-dose 25(OH)D
  Arms: Vitamin D3 6000 IU
Drug: Vitamin D3 400 IU — Subjects will receive 400 IU/day of vitamin D3 daily by mouth.
  Other Names: standard-dose vitamin D; standard-dose cholecalciferol (D3); standard-dose 25(OH)D
  Arms: Vitamin D3 400 IU

SUMMARY:
The primary objective of this study is to evaluate the effects of 18 weeks of high-dose vitamin D3 supplementation compared with standard-dose vitamin D3 supplementation on immune function, glucose homeostasis, and bone metabolism in children with systemic lupus erythematosus (SLE) and serum 25-hydroxyvitamin D [25(OH)D] levels ≤20 ng/mL.

DETAILED DESCRIPTION:
This is a multi-center, phase II, 18-week, two arm, unblinded randomized clinical trial.

Seventy-eight pediatric subjects with SLE and 25(OH)D levels ≤ 20 ng/mL will be randomized in a 1:1 ratio to receive either standard-dose (400 IU/day) or high-dose (6,000 IU/day) vitamin D3 for 18 weeks based upon weight at baseline. Subjects randomized to the high-dose vitamin D3 treatment arm will receive 6,000 IU per day from baseline until the subject's vitamin D levels reach ≥ 40 ng/mL at which point the vitamin D3 dose will be reduced to 4,000 IU per day. Subjects randomized to the high-dose treatment arm weighing < 40 kg will receive supplementation five days per week and all other subjects will receive supplementation seven days a week.

In addition to the baseline, and weeks 6, 12, and 18 visits, subjects randomized to the high-dose treatment arm will return at Weeks 3 and 9 to assess for symptoms of vitamin D toxicity. If a subject in the high-dose arm is found to exhibit evidence of vitamin D toxicity at the week 12 visit, he/she will be asked to return to their clinical research site for an additional vitamin D toxicity assessment at week 15. Study personnel will record each subject's interval history, assess adverse events, disease activity, and collect samples for safety and mechanistic assessments.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed by the subject or parent/guardian as appropriate; child assent as appropriate;
* Before the age of 19, met at least 4 of the 11 modified American College of Rheumatology (ACR) 1982 Revised Criteria for the Classification of Systemic Lupus Erythematosus as updated in 1997;
* Date of SLE diagnosis (as described in Inclusion Criterion 2) at least 24 weeks prior to randomization;
* Serum 25-hydroxyvitamin D [25(OH)D] < 20 ng/mL at Screening;
* SELENA SLEDAI score > 0 and < 8 at Screening and at Baseline;
* If taking prednisone (or equivalent corticosteroid), the dose must be ≤ 15 mg/day or ≤0.5 mg/kg/day, whichever is lower, and stable for at least four weeks prior to randomization. Note, if subjects are taking steroids every other day, divide their dose by 2 to evaluate eligibility;
* Stable immunosuppressive dose for at least 12 weeks prior to randomization;

  --Immunosuppressive medications allowed include mycophenolate (MMF), azathioprine, methotrexate, antimalarial medications (e.g., hydroxychloroquine), cyclosporine A (CsA), tacrolimus, intravenous immune globulin (IVIG), and abatacept.
* Body weight > 25 kg;
* Able to swallow pills;
* Males and females with reproductive potential must agree to practice effective measures of birth control.

Exclusion Criteria:

* Any condition or treatment that, in the opinion of the investigator, places the subject at an unacceptable risk as a participant in the trial;
* Current pharmacologic vitamin D2 or D3 intake > 800 IU daily or use of calcitriol at any dose over the past four weeks prior to randomization;
* Cyclophosphamide or IV glucocorticoid exposure within 12 weeks prior to randomization;
* Any BILAG A or B manifestation with the exception of a BILAG B mucocutaneous manifestation at screening, and excluding the renal BILAG criteria (see rituximab or belimumab criterion, below);
* Significant renal insufficiency defined as:

  * Estimated GFR < 60 mL/min/1.73m^2 or estimated GFR < 90 mL/min/1.73m^2 with a reduction of the GFR by > 15% from the last measurement;
  * Urine dipstick value of 2+ or higher for protein, unless this is a stable value from the last measurement or, urine protein-creatinine ratio ≥ 50 mg/mmol unless the value represents an improvement of ≥ 25% from the last measurement.
* Rituximab or belimumab exposure use within 24 weeks prior to randomization;
* The following laboratory parameters at the Screening visit:

  * Platelets < 50,000; WBC < 2,500; ANC < 1,000;
  * Hemoglobin < 9 mg/dL;
  * ALT, AST, bilirubin > 2x upper limit of normal (ULN);
  * Hypercalcemia (calcium > ULN);
  * Hypercalciuria (urinary calcium/creatinine ratio > 0.2).
* Primary hyperparathyroidism (known);
* History of nephrolithiasis (known);
* Diabetes mellitus requiring insulin therapy;
* Medications that interfere with vitamin D absorption;
* History of vertebral compression fractures (known);
* Pregnancy (girls ≥ 11 years of age must have a negative urine/serum pregnancy test);
* A history of non-adherence/non-compliance;
* Other investigational drug and/or treatment during the four weeks or seven half-lives of the other investigational drug prior to the start of study product dosing (Day 0), whichever is the greater length of time to enrollment;
* Current diagnosis of cancer or chronic infection such as Hepatitis B, Hepatitis C, or tuberculosis;
* Treatment with digoxin;
* Flu (influenza) vaccination within one week prior to randomization.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon M Burnham, MD, MSCE, Study Chair — University of Pennsylvania; Emily Von Scheven, MD, MAS, Study Chair — University of California, San Francisco
Locations (13):
- United States (13):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital, Stanford University, Palo Alto, California
  - UCSF School of Medicine, San Francisco, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D3 6000 IU: Participants received an 18-week course of oral Vitamin D3 (cholecalciferol, 6,000 international units [IU] daily).
- Vitamin D3 400 IU: Participants received an 18-week course of oral Vitamin D3 (cholecalciferol, 400 international units [IU] daily).
Period: Overall Study
Arm/Group | Vitamin D3 6000 IU | Vitamin D3 400 IU
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The population included all subjects who were randomized to receive either Vitamin D3 6000 IU daily or 400 IU daily.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 6000 IU | Vitamin D3 400 IU | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.3 (3.8) | 13.5 (0.6) | 14.7 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7
25(OH)D at Screening [Mean (Standard Deviation); unit: ng/mL] — 25(OH)D is also called vitamin D3. Participants were required to have a screening value of less than 20 ng/mL to be eligible for the study.
  ng/mL | 9.3 (3.9) | 16.1 (2.5) | 13.2 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Average IFN Module Expression Level
Description: No mechanistic analyses were performed due to recruitment feasibility issues.
Time Frame: Baseline to Week 18
Population: Data were not collected and therefore no analyses could be performed.
Arm/Group | Vitamin D3 6000 IU | Vitamin D3 400 IU
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Percentage of Subjects by Treatment Arm Experiencing Any Adverse Event (AE) ≥ Grade 3
Description: Adverse event grading based on National Cancer Institute- Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.0
Time Frame: Baseline to 18 Weeks
Population: Intent-to-treat
Measure: Number; unit: Percentage of Participants
Arm/Group | Vitamin D3 6000 IU | Vitamin D3 400 IU
Number analyzed (Participants) | 3 | 4
Percentage of Participants | 0 | 25

ADVERSE EVENTS:
Time Frame: From the time of administration of the first dose of study drug until the participant completed study participation, an average of 18 weeks.
Arm/Group | Vitamin D3 6000 IU | Vitamin D3 400 IU
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/3 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D3 6000 IU (N=3) | Vitamin D3 400 IU (N=4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hypercalciuria (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study terminated early due to recruitment feasibility issues. Seven subjects were enrolled and received treatment in contrast to the planned number of 78 subjects for randomization/receipt of treatment. No mechanistic analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No